CLINICAL TRIAL: NCT02319538
Title: Surgical Treatment of Hashimotos Disease. Effect on Antibodies and Clinical Symptoms.
Brief Title: Hashimoto - a Surgical Disease. Total Thyroidectomy Makes Antibodies Disappear and Ameliorates Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Helse Stavanger HF (Other Government); Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Ivar Guldvog, Consultant, Sykehuset Telemark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DTG 031100-031230
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Hashimoto's Disease
Keywords: Chronic thyroiditis; Total thyroidectomy; Anti-TPO; PROMs; SF36; Fatigue questionnaire; Fatigue; Autoimmune symptoms; HADs; FSS; fVAS
MeSH Terms: conditions — Hashimoto Disease; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-surgical treatment only (No Intervention): Control arm. This arm receives standard medical hormone treatment (Thyroxine substitution) only and no surgical intervention.
- Total thyroidectomy performed (Active Comparator): Surgical arm.The approach for total thyroidectomy will be a complete removal of all visible, and immunological active thyroid tissue with a high accuracy, with a special focus on three sites; 1) The angle where the recurrent laryngeal nerve enters the cricothyroid membrane, 2) The pyramidal lobe and 3) The hilus where the superior vessels are entering the field. Standard Thyroxine supplementation maintained as in the control group.
  Interventions: Procedure: Total thyroidectomy performed

INTERVENTIONS:
Procedure: Total thyroidectomy performed — Surgery combined with standard thyroxine treatment
  Arms: Total thyroidectomy performed

SUMMARY:
The investigators have already proven that absolute total thyroidectomy gives elimination of anti-TPO antibodies. Our hypothesis is that this elimination also eliminates the typical Hashimoto symptoms, namely: Serious tiredness, increased need of sleep, pain in musculature and joints and dryness in eyes and mouth. The prerequisite for this effect is that the total thyroidectomy is meticulously performed. There exists no other treatment that can eliminate the antibodies. The study is randomized between operation and ordinary conservative medical treatment with thyroxine control and supplementation. The symptoms in both groups are evaluated by 5 different Quality of Life schemes, internationally approved.

DETAILED DESCRIPTION:
The study hypothesis is that elimination of anti-TPO antibodies ameliorates the typical Hashimoto symptoms like tiredness,increased need of sleep, pain in musculature and joints and dryness in eyes and mouth. It is necessary that the total thyroidectomy is meticulously performed. We have proven the effect on the antibodies, and we have also proven that the operation procedure can be performed without more complications like recurrent nerve damage and hypocalcemia. Neutrality is secured by randomization done by a neutral institution, laryngoscopy by neutral doctors and instructions filling out the QoL-schemes performed by non-biased study nurses.

The study runs for at least 18 months with controls every 6 months. Blood samples are taken and international approved QoL-schemes are filled in. In addition to the randomised main group a side group of patients fulfilling 2 of the 3 inclusion criteria are followed in parallel in order to elucidate the spontaneous development of the disease and showing critical values of antibodies making the symptoms turn up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred due to typical symptoms, believed to be related to Hashimoto´s disease, but not relieved by thyroxin substitution. Optimal thyroid substitution treatment is already provided.
2. Anti-TPO>1000
3. Hypothyroidism with a need for thyroxin supplementation
4. Written informed consent by the patient - information particularly emphasising and quantifying the risk of complications (e.g. recurrent laryngeal nerve palsy). The patient should be informed by a medical endocrinologist as well as a surgeon.

Exclusion Criteria:

1. Patients <18 years of age.
2. Pregnancy.
3. Unable to comprehend information adequately to give informed consent.
4. General anaesthesiological contraindications.
5. An unexpected finding of cancer in the surgical group is not a reason for exclusion per se, but this group should be analyzed separately. It is expected that any different loading in Quality of life would bias the medically treated group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-02-13 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Better outcome in Quality of Life by operation | 18 months
  The patiens are followed for 18 months with blood samples and filling in Quality of Life schemes every 6 months

SECONDARY OUTCOMES:
Lowering of antibodies (Blood samples) | 18 months
  Blood samples every 6 months

OTHER OUTCOMES:
Safety in performing absolute total thyroidectomy (recurrence nerve and long lasting hypocalcemia) | 12 months
  Safety concerning the recurrence nerve and long lasting hypocalcemia. Interim analysis after 75 patients.
Interim analysis after 75 patients concerning safety (recurrent nerve control by laryngoscopy and hypocalcemia control by blood samples) | 12 months
  The patients operated upon are investigated after 12 months concerning safety. The recurrent nerve control by laryngoscopy and hypocalcemia control by blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Ivar Guldvog, MD, PhD, Principal Investigator — Sykehuset Telemark; Hege Kersten, PhD, Study Director — Sykehuset Telemark
Locations (1):
- Telemark Hospital Trust, surgical department, Skien, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guldvog I, Reitsma LC, Johnsen L, Lauzike A, Gibbs C, Carlsen E, Lende TH, Narvestad JK, Omdal R, Kvaloy JT, Hoff G, Bernklev T, Soiland H. Thyroidectomy Versus Medical Management for Euthyroid Patients With Hashimoto Disease and Persisting Symptoms: A Randomized Trial. Ann Intern Med. 2019 Apr 2;170(7):453-464. doi: 10.7326/M18-0284. Epub 2019 Mar 12. PMID 30856652